CLINICAL TRIAL: NCT02143947
Title: The Effect of Two Different Custom Molded Foot Orthoses on Inter-segmental Foot Kinematics and the EMG Activity of Selected Lower Leg Muscles During Walking and Running.
Brief Title: Custom Molded Foot Orthoses Effect on Foot Kinematics and Lower Extremity Electromyography During Walking and Running.
Acronym: SOLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quinnipiac University (Other)
Collaborators: Sole Supports, Inc (Unknown)
Responsible Party: Principal Investigator, Juan C. Garbalosa, PT, PhD, Director, Motion Analysis Laboratory, Clinical Associate Proffessor of Physical Therapy, Quinnipiac University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HEC 1404
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-04

CONDITIONS: Lower Extremity Pain of a Mechanical Origin
Keywords: Orthoses; Foot; Kinematics; EMG; Biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full Contact Orthosis (Experimental): Full Contact Orthosis
  Interventions: Device: Full Contact Orthosis
- Maximal Arch Subtalar Stabilization (Experimental): Maximal Arch Subtalar Stabilization Orthoses
  Interventions: Device: Maximal Arch Subtalar Stabilization

INTERVENTIONS:
Device: Maximal Arch Subtalar Stabilization — Custom made semi-rigid thermoplastic heel cup extending to the base of the metatarsals with a full foot length 3.0mm thick EVA and ultra-suede top cover
  Arms: Maximal Arch Subtalar Stabilization
Device: Full Contact Orthosis — The Full Contact orthosis is constructed from a 5/32" blue polypropylene with posting material comprised of white polypropylene.
  Arms: Full Contact Orthosis

SUMMARY:
The purpose of this study was to determine the effectiveness of two types of in-shoe custom made orthotics in altering the motion of the foot and muscle activity of select muscles of the lower leg in individuals experiencing lower extremity symptoms of a non traumatic origin. We hypothesized that orthotics would decrease the extent of motion of the during walking and running when compared to a barefoot condition. The investigators further hypothesized that orthotics would decrease the amount of muscle activity seen during walking and running when compared to barefoot walking.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have complaints of lower extremity or foot pain of a non-traumatic, mechanical origin.
* Subjects must have at least 60 degrees of frontal plane forefoot on rearfoot passive range of motion (as determined by a modified Gib test in the symptomatic lower extremity.
* Subjects must be able to walk independently on a treadmill at a speed of 4.8 kmh.
* Subjects must have been referred by a health care professional for an orthosis fitting.

Exclusion Criteria:

* Subjects having less than 60 degrees of forefoot on rearfoot frontal plane passive range of motion.
* Subjects having a history of a fracture of the foot or ankle.
* Subjects having any previous illness, surgery or other characteristic (e.g., cardiovascular, musculoskeletal or neuromuscular problems) that would affect their lower extremity function or ability to walk independently.
* Subjects having knee, lower leg or foot pain of a non-mechanical nature.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Garbalosa, PT, PhD, Principal Investigator — Quinnipiac University
Locations (1):
- Motion Analysis Laboratory, Quinnipiac Unviersity, Hamden, Connecticut, United States

REFERENCES:
- [Derived] Garbalosa JC, Elliott B, Feinn R, Wedge R. The effect of orthotics on intersegmental foot kinematics and the EMG activity of select lower leg muscles. Foot (Edinb). 2015 Dec;25(4):206-14. doi: 10.1016/j.foot.2015.07.005. Epub 2015 Jul 14. PMID 26362236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A convenience sample of subjects was obtained via email and bulletin board postings at a local private university. Recruitment commenced 9/1/08 and ended on 2/1/09.
Pre-assignment Details: There were no significant events associated with this study.
Groups:
- Full Contact Orthosis: Full Contact Orthosis
  Full Contact Orthosis: The full contact in-shoe orthosis is constructed from a 5/32" blue polypropylene with posting material comprised of white polypropylene.
- Maximal Arch Subtalar Stabilization: Maximal Arch Subtalar Stabilization Orthoses
  Maximal Arch Subtalar Stabilization: The in-shoe orthosis is a custom made semi-rigid thermoplastic heel cup extending to the base of the metatarsals with a full foot length 3.0mm thick EVA and ultra-suede top cover
Period: Overall Study
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Started | 36 | 44
Completed | 32 | 42
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Population: The number participants for analysis was based upon the number of participants who attended the first data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization | Total
Number analyzed (Participants) | 36 | 44 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.7 (6.6) | 20.3 (1.5) | 20.9 (4.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 4 | 11
  Between 18 and 65 years | 29 | 40 | 69
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 36 | 44 | 80
Region of Enrollment [Number; unit: participants]
  United States | 36 | 44 | 80
Visual Analogue Pain Scale [Mean (Standard Deviation); unit: units on a scale] — The visual analogue scale has a range from 0 to 10. 0 representing no pain, 10 representing the worse possible pain. Higher scores are considered worse.
  units on a scale | 7.2 (1.7) | 7.0 (2.0) | 7.0 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Rearfoot Eversion Motion During Stance
Description: The rearfoot eversion motion during the stance phase of walking with the subject wearing a sandal and their assigned orthotic (Full Contact or Maximal Arch Subtalar Stabilization) was recorded 5 weeks post receiving their assigned orthotic. The stance phase of walking was divided into 4 subphases (Phase 1: 0 to 17%, Phase 2: 18 to 50%, Phase 3: 51 to 83%, and Phase 3: 84 to 100% of stance) and the maximum rearfoot eversion during each subphase determined.
Time Frame: Absolute values measured at 5 weeks
Population: The number of participants used for the analysis was based upon the availability of complete data sets.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Number analyzed (Participants) | 26 | 26
Degrees
  Sandal Only, Phase 1 | 1.1 (9.9) | 1.1 (11.3)
  Sandal Only, Phase 2 | 2.9 (10.0) | 3.0 (10.3)
  Sandal Only, Phase 3 | 2.2 (9.2) | 2.7 (9.2)
  Sandal Only, Phase 4 | -2.4 (7.5) | -1.1 (8.8)
  Sandal-Orthotic Only, Phase 1 | 0.2 (9.9) | 1.7 (11.5)
  Sandal-Orthotic Only, Phase 2 | 1.3 (9.6) | 3.1 (10.5)
  Sandal-Orthotic Only, Phase 3 | 1.3 (9.2) | 2.7 (9.9)
  Sandal-Orthotic Only, Phase 4 | -2.7 (8.1) | -0.9 (9.2)
Statistical Analysis 1: Comparison: Full Contact Orthosis vs Maximal Arch Subtalar Stabilization; Test type: Superiority or Other; p > .10, Mixed Models Analysis

2. Secondary Outcome: Maximum Electromyographic Activity of Lower Leg Muscles
Description: The maximum electromyographic activity of the lower leg muscles is with respect to the barefoot condition. The electromyographic activity of the lower extremity muscles were recorded during the stance phase of walking while barefoot and while wearing their assigned orthotic (Full Contact or Maximal Arch Subtalar Stabilization). All electromyographic measurements were taken at the 5 week time point. The peak electromyographic activity during the stance phase of barefoot walking was determined. The electromyographic activity during the orthotic condition was amplitude normalized to the barefoot condition by dividing the electromyographic activity of the orthotic condition by the peak barefoot electromyographic activity and multiplying by 100. The stance phase of walking was then divided into 4 subphases (Phase 1: 0 to 17%, Phase 2: 18 to 50%, Phase 3: 51 to 83%, and Phase 3: 84 to 100% of stance) and the peak amplitude normalized electromyographic activity of each subphase det
Time Frame: Absolute values measured at 5 weeks
Population: The number of participants used for the analysis was based upon the availability of complete data sets.
Measure: Mean (Standard Deviation); unit: percentage of maximum electromyo actvity
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Number analyzed (Participants) | 26 | 26
percentage of maximum electromyo actvity
  Tibialis Anterior Phase 1 | 69.5 (24.8) | 71.2 (21.9)
  Tibailis Anterior Phase 2 | 23.6 (14.1) | 27.1 (23.6)
  Tibialis Anterior Phase 3 | 29.6 (14.9) | 30.9 (19.7)
  Tibialis Anterior Phase 4 | 41.9 (14.4) | 46.8 (16.7)
  Tibialis Posterior Phase 1 | 45.5 (32.8) | 50.2 (29.7)
  Tibialis Posterior Phase 2 | 35.1 (26.6) | 46.0 (28.4)
  Tibialis Posterior Phase 3 | 49.4 (48.6) | 53.1 (35.2)
  Tibialis Posterior Phase 4 | 27.4 (48.7) | 20.9 (19.6)
  Peroneus Longus Phase 1 | 41.5 (29.2) | 40.8 (24.4)
  Peroneus Longus Phase 2 | 48.1 (33.5) | 58.7 (37.5)
  Peroneus Longus Phase 3 | 52.5 (35.1) | 55.7 (36.9)
  Peroneus Longus Phase 4 | 18.8 (18.6) | 25.8 (28.6)
Statistical Analysis 1: Comparison: Full Contact Orthosis vs Maximal Arch Subtalar Stabilization; Test type: Superiority or Other; p = .036, Mixed Models Analysis

3. Secondary Outcome: Maximum Forefoot Inversion During Stance
Description: The forefoot inversion motion during the stance phase of walking with the subject wearing a sandal and their assigned orthotic (Full Contact or Maximal Arch Subtalar Stabilization) was recorded 5 weeks post receiving their assigned orthotic. The stance phase of walking was divided into 4 subphases (Phase 1: 0 to 17%, Phase 2: 18 to 50%, Phase 3: 51 to 83%, and Phase 3: 84 to 100% of stance) and the maximum forefoot inversion during each subphase determined.
Time Frame: Absolute values measured at 5 weeks
Population: The number of participants used for the analysis was based upon the availability of complete data sets.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Number analyzed (Participants) | 26 | 26
Degrees
  Sandal Only, Phase 1 | -13.0 (9.7) | -13.8 (12.2)
  Sandal Only, Phase 2 | -12.2 (10.2) | -12.9 (11.8)
  Sandal Only, Phase 3 | -12.7 (8.9) | -14.0 (10.2)
  Sandal Only, Phase 4 | -12.7 (8.5) | -14.7 (10.9)
  Sandal-Orthotic Only, Phase 1 | -12.0 (10.5) | -14.2 (12.0)
  Sandal-Orthotic Only, Phase 2 | -11.4 (10.8) | -13.6 (11.7)
  Sandal-Orthotic Only, Phase 3 | -12.6 (9.8) | -14.0 (10.7)
  Sandal-Orthotic Only, Phase 4 | -11.9 (9.3) | -14.6 (11.0)
Statistical Analysis 1: Comparison: Full Contact Orthosis vs Maximal Arch Subtalar Stabilization; Test type: Superiority or Other; p > .10, Mixed Models Analysis

4. Secondary Outcome: Maximum First Ray Complex Plantarflexion During Stance
Description: The first ray complex plantarflexion during the stance phase of walking with the subject wearing a sandal and their assigned orthotic (Full Contact or Maximal Arch Subtalar Stabilization) was recorded 5 weeks post receiving their assigned orthotic. The stance phase of walking was divided into 4 subphases (Phase 1: 0 to 17%, Phase 2: 18 to 50%, Phase 3: 51 to 83%, and Phase 3: 84 to 100% of stance) and the maximum first ray complex plantarflexion during each subphase determined.
Time Frame: Absolute values measured at 5 weeks
Population: The number of participants used for the analysis was based upon the availability of complete data sets.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Number analyzed (Participants) | 26 | 26
Degrees
  Sandal Only, Phase 1 | -6.96 (3.8) | -4.95 (5.0)
  Sandal Only, Phase 2 | -3.37 (3.3) | -1.22 (4.8)
  Sandal Only, Phase 3 | -1.25 (2.9) | 1.54 (5.3)
  Sandal Only, Phase 4 | -4.07 (4.4) | -4.39 (6.0)
  Sandal-Orthotic, Phase 1 | -6.49 (3.8) | -4.67 (4.4)
  Sandal-Orthotic, Phase 2 | -2.92 (3.3) | -1.5 (4.2)
  Sandal-Orthotic, Phase 3 | -1.03 (2.9) | .62 (4.4)
  Sandal-Orthotic, Phase 4 | -4.07 (4.4) | -3.24 (5.4)
Statistical Analysis 1: Comparison: Full Contact Orthosis vs Maximal Arch Subtalar Stabilization; Test type: Superiority or Other; p < .05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for one year
Description: Adverse event information was collected at the time of the 5 week data collection via direct observation and a 3 and 6 month and 1 year follow up via telephone or email interview.
Arm/Group | Full Contact Orthosis | Maximal Arch Subtalar Stabilization
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/44
Other Adverse Events (participants affected / at risk) | 0/36 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No